CLINICAL TRIAL: NCT03629860
Title: Assessment of Mandibular Ascending Ramus Cortical Plates for Reconstruction of Atrophic Maxillary Ridges Versus Chin Cortical Plates(Randomized Clinical Tial)
Brief Title: Ascending Ramus Versus Chin Cortical Plates for Reconstruction of Atrophic Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed yousri said zayed, B.D.S,Principal investigator,dentist, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Ahmed yousri
Record Dates: First submitted 2018-08-06; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Atrophy of Edentulous Maxillary Alveolar Ridge
Keywords: Atrophic, augmetation, bone regeneration
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Intervention Model Description: Assessment of ascending ramus cortical plate for reconstruction of atrophic maxillary ridges versus chin cortical plates (Randomized clinical trial)
Who Masked: Participant
Masking Description: Assessment of ascending ramus cortical plate for reconstruction of atrophic maxillary ridges versus chin cortical plates (Randomized clinical trial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ascending ramus group (Active Comparator): * Local anesthesia will be given to the patient
  * flap will be reflected to expose the facial wall of the maxilla then The ascending ramus is accessed.
  * A disc bur will be used to make a rectangular osteotomy
  * The block bone graft is removed from ascending ramus to recipient site the fixed by mini screws
  * Doner site flap is closed by using interrupted internal sutures.
  * after atrophic maxillary alveolar ridge augmentation,sub mucosal periosteal releasing cuts is done
  * Post-operative medications will be prescribed as follows: amoxicillin/clavulanic acid tablets 10mg/kg every 12 hours for 7 days, metronidazole 5 mg/kg every 8 hours for 7 days
  Interventions: Procedure: Atrophic maxillary alveolar ridge augmentation
- Chin Group (Active Comparator): * Local anesthesia will be given to the patient
  * flap will be reflected to expose the facial wall of the maxilla then The chin is accessed.
  * A disc bur will be used to make a rectangular osteotomy
  * The block bone graft is removed from chin to recipient site the fixed by mini screws
  * Doner site flap is closed by using interrupted internal sutures
  * after atrophic maxillary alveolar ridge augmentation,submucosal periosteal releasing cuts is done
  * Post-operative medications will be prescribed as follows: amoxicillin/clavulanic acid tablets 10mg/kg every 12 hours for 7 days, metronidazole 5 mg/kg every 8 hours for 7days
  Interventions: Procedure: Atrophic maxillary alveolar ridge augmentation

INTERVENTIONS:
Procedure: Atrophic maxillary alveolar ridge augmentation — Autogenous bone blocks from chin and ascending ramus are obtained and used for reconstruction of atrophic maxillary ridges

SUMMARY:
Assessment of ascending ramus cortical plate for reconstruction of atrophic maxillary ridges versus chin cortical plates (Randomized clinical trial)

DETAILED DESCRIPTION:
Assessment of ascending ramus cortical plate for reconstruction of atrophic maxillary ridges versus chin cortical plates (Randomized clinical trial) To know what is better and more efficient chin or ascending ramus cortical plates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophic maxilla with residual bone height from 3 to 4mm.
* Both sexes

Exclusion Criteria:

* Intraoral soft and hard tissue pathology.
* Systemic condition that contraindicate implant basement.
* Psychiatric problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-02-08 (Estimated); Study Completion 2019-04-09 (Estimated)

PRIMARY OUTCOMES:
width and height of the bone gained by the procedure and the new measures from a physiologic vital structures e.g( nasal floor, maxillary sinus or even occlusal plan) | 6 months
  new bone formation

SECONDARY OUTCOMES:
Histomorphometric analysis bone area percent | 6 months
  Nature and quality of new bone histology

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Yousri, Bsd, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Al-Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Websites and papers

REFERENCES:
- [Background] Ali SA, Karthigeyan S, Deivanai M, Kumar A. Implant rehabilitation for atrophic maxilla: a review. J Indian Prosthodont Soc. 2014 Sep;14(3):196-207. doi: 10.1007/s13191-014-0360-4. Epub 2014 Apr 22. PMID 25183902
- [Background] Sorni M, Guarinos J, Garcia O, Penarrocha M. Implant rehabilitation of the atrophic upper jaw: a review of the literature since 1999. Med Oral Patol Oral Cir Bucal. 2005 Apr 1;10 Suppl 1:E45-56. English, Spanish. PMID 15800467
- [Background] Dym H, Huang D, Stern A. Alveolar bone grafting and reconstruction procedures prior to implant placement. Dent Clin North Am. 2012 Jan;56(1):209-18, x. doi: 10.1016/j.cden.2011.09.005. PMID 22117951
- [Background] Bellini CM, Romeo D, Galbusera F, Agliardi E, Pietrabissa R, Zampelis A, Francetti L. A finite element analysis of tilted versus nontilted implant configurations in the edentulous maxilla. Int J Prosthodont. 2009 Mar-Apr;22(2):155-7. PMID 19418861
- [Background] Bidra AS, Almas K. Mini implants for definitive prosthodontic treatment: a systematic review. J Prosthet Dent. 2013 Mar;109(3):156-64. doi: 10.1016/S0022-3913(13)60035-9. PMID 23522364
- [Background] Chiriac G, Herten M, Schwarz F, Rothamel D, Becker J. Autogenous bone chips: influence of a new piezoelectric device (Piezosurgery) on chip morphology, cell viability and differentiation. J Clin Periodontol. 2005 Sep;32(9):994-9. doi: 10.1111/j.1600-051X.2005.00809.x. PMID 16104964
- [Background] Enneking WF, Eady JL, Burchardt H. Autogenous cortical bone grafts in the reconstruction of segmental skeletal defects. J Bone Joint Surg Am. 1980 Oct;62(7):1039-58. PMID 7000788
- [Background] Menini M, Signori A, Tealdo T, Bevilacqua M, Pera F, Ravera G, Pera P. Tilted implants in the immediate loading rehabilitation of the maxilla: a systematic review. J Dent Res. 2012 Sep;91(9):821-7. doi: 10.1177/0022034512455802. Epub 2012 Jul 31. PMID 22851285
- [Background] Peleg M, Mazor Z, Garg AK. Augmentation grafting of the maxillary sinus and simultaneous implant placement in patients with 3 to 5 mm of residual alveolar bone height. Int J Oral Maxillofac Implants. 1999 Jul-Aug;14(4):549-56. PMID 10453671
- [Background] Topolovec-Vranic J, Canzian S, Innis J, Pollmann-Mudryj MA, McFarlan AW, Baker AJ. Patient satisfaction and documentation of pain assessments and management after implementing the adult nonverbal pain scale. Am J Crit Care. 2010 Jul;19(4):345-54; quiz 355. doi: 10.4037/ajcc2010247. PMID 20595216